CLINICAL TRIAL: NCT03715933
Title: An Open-Label, Multicenter, First-in-Human, Phase 1 Dose-Escalation and Multicohort Expansion Study of INBRX-109 in Subjects With Locally Advanced or Metastatic Solid Tumors Including Sarcomas
Brief Title: Phase 1 Study of INBRX-109 in Subjects With Locally Advanced or Metastatic Solid Tumors Including Sarcomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Inhibrx Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ph1 INBRX-109
Record Dates: First submitted 2018-10-11; First posted 2018-10-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Ewing Sarcoma
Keywords: Phase 1; Phase 1 Clinical Trial; Solid Tumors; Sarcoma; DR5; Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Sarcoma | interventions — Irinotecan; Temozolomide; Carboplatin; Pemetrexed; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Dose Escalation (Complete) (Experimental): INBRX-109 will be escalated (3+3 design) in subjects with locally advanced or metastatic solid tumors including sarcomas.
  Interventions: Drug: INBRX-109
- Expansion Malignant Pleural Mesothelioma (Complete) (Experimental): Subjects with malignant pleural mesothelioma will be treated with single-agent INBRX-109 at either the MTD or RP2D.
  Interventions: Drug: INBRX-109
- Expansion Gastric Adenocarcinoma (Complete) (Experimental): Subjects with gastric adenocarcinoma will be treated with single-agent INBRX-109 at either the MTD or RP2D.
  Interventions: Drug: INBRX-109
- Expansion Colorectal Adenocarcinoma (Complete) (Experimental): Subjects with colorectal (CRC) adenocarcinoma will be treated with single-agent INBRX-109 at either the MTD or RP2D.
  Interventions: Drug: INBRX-109
- Expansion Sarcomas (Complete) (Experimental): Subjects with certain sarcoma subtypes will be treated with single-agent INBRX-109 at either the MTD or RP2D.
  Interventions: Drug: INBRX-109
- Combination Expansion Malignant Pleural Mesothelioma (Complete) (Experimental): Subjects with malignant pleural mesothelioma will be treated with INBRX-109 in combination with chemotherapies (carboplatin, cisplatin, carboplatin and pemetrexed, or cisplatin and pemetrexed)
  Interventions: Drug: INBRX-109; Drug: carboplatin; Drug: pemetrexed
- Combination Expansion Pancreatic Adenocarcinoma (Complete) (Experimental): Subjects with pancreatic adenocarcinoma will be treated with INBRX-109 in combination with 5FU/irinotecan based chemotherapy
  Interventions: Drug: INBRX-109; Drug: Irinotecan; Drug: Leucovorin; Drug: Fluorouracil
- Combination Expansion Ewing Sarcoma (Experimental): Subjects with Ewing Sarcoma will be treated with INBRX-109 in combination with irinotecan and temozolomide
  Interventions: Drug: INBRX-109; Drug: Irinotecan; Drug: Temozolomide
- Combination Expansion Colorectal Adenocarcinoma (Complete) (Experimental): Subjects with colorectal adenocarcinoma will be treated with INBRX-109 in combination with FOLFIRI based chemotherapy
  Interventions: Drug: INBRX-109; Drug: Irinotecan; Drug: Leucovorin; Drug: Fluorouracil
- Expansion Solid Tumors (Complete) (Experimental): Subjects with Solid tumors and high BMI will be treated with single-agent INBRX-109 at either the MTD or RP2D.
  Interventions: Drug: INBRX-109
- Combination Expansion SDH-deficient solid tumors or GIST (Complete) (Experimental): Subjects with SDH-deficient solid tumors or GIST will be treated with INBRX-109 in combination with temozolomide
  Interventions: Drug: INBRX-109; Drug: Temozolomide

INTERVENTIONS:
Drug: INBRX-109 — Tetravalent DR5 Agonist Antibody
Drug: Irinotecan — Chemotherapy
  Arms: Combination Expansion Colorectal Adenocarcinoma (Complete); Combination Expansion Ewing Sarcoma; Combination Expansion Pancreatic Adenocarcinoma (Complete)
Drug: Temozolomide — Chemotherapy
  Arms: Combination Expansion Ewing Sarcoma; Combination Expansion SDH-deficient solid tumors or GIST (Complete)
Drug: carboplatin — chemotherapy
  Arms: Combination Expansion Malignant Pleural Mesothelioma (Complete)
Drug: pemetrexed — chemotherapy
  Arms: Combination Expansion Malignant Pleural Mesothelioma (Complete)
Drug: Leucovorin — chemotherapy
  Arms: Combination Expansion Colorectal Adenocarcinoma (Complete); Combination Expansion Pancreatic Adenocarcinoma (Complete)
Drug: Fluorouracil — chemotherapy
  Arms: Combination Expansion Colorectal Adenocarcinoma (Complete); Combination Expansion Pancreatic Adenocarcinoma (Complete)

SUMMARY:
This is a first-in-human, open-label, non-randomized, three-part phase 1 trial of INBRX-109, which is a recombinant humanized tetravalent antibody targeting the human death receptor 5 (DR5).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥12 to less than 85 years for Ewing sarcoma and 18 to less than 85 years of age for other tumors.
2. Part 3 combination therapy expansion tumor types:

   * Histologically confirmed Ewing sarcoma with a classical fusion: Patients with locally advanced or metastatic, unresectable, relapsed, or refractory disease who have received at least 1 but no more than 2 prior lines of systemic treatment with a preferred first line chemotherapy regimens.
   * Colorectal adenocarcinoma: Patients with locally advanced or metastatic, unresectable disease, who have received at least 2 but no more than 3 prior lines of systemic therapy.
3. Measurable disease as defined by RECISTv1.1 (or modified RECIST for mesothelioma) criteria.
4. Adequate hematologic, coagulation, hepatic and renal function as defined per protocol.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1, or Karnofsky Performance Status score of ≥60, or Lansky Play-Performance Scale for Children score ≥60 (for patients less than 16 years).
6. Estimated life expectancy of at least 12 weeks.
7. Availability of archival tissue or fresh cancer biopsy are mandatory.

Exclusion Criteria:

1. Prior treatment with or exposure to DR5 agonists.
2. Receipt of any anticancer therapy (including investigational agents) within 4 weeks or within 5 half-lives prior to the first dose of study treatment. Exceptions per protocol.
3. Allergy or sensitivity to INBRX-109 or known allergies to CHO-produced antibodies.
4. Receipt of radiotherapy within 4 weeks prior to the first dose of study treatment, and liver-directed within 12 months prior to the first dose of study drug.
5. Subject has undergone allogeneic hematopoietic stem cell or bone marrow transplantation within the last 5 years. Exceptions per protocol.
6. Prior or concurrent malignancies. Exceptions per protocol.
7. Hematologic malignancies.
8. Symptomatic active primary CNS tumors, leptomeningeal disease, and CNS metastases. Exceptions per protocol. Patients with any evidence or history of multiple sclerosis (MS) or other demyelinating disorders are excluded.
9. Chronic liver diseases including fatty liver. Exception: Patients < 45 years old with fatty liver disease may be accepted as long as adequate hepatic function as defined in the inclusion/exclusion criteria is confirmed.
10. Acute viral or toxic liver disease within 12 months prior to the first dose of study drug.
11. Evidence or history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection.
12. Known sensitivity or contraindications to the following drugs:

    * Ewing sarcoma: irinotecan or TMZ
    * colorectal adenocarcinoma: FU, leucovorin, or irinotecan
13. Clinically significant cardiac condition, including myocardial infarction, uncontrolled angina, cerebrovascular accident, or other acute uncontrolled heart disease less than 3 months prior to enrollment.
14. Acute, hemodynamically significant deep vein thrombosis or clinically significant pulmonary embolism not resolved or stable for at least 3 months prior to the start of study treatment.
15. Major surgery within 4 weeks prior to enrollment on this trial.
16. Systemic infection requiring antibiotics within 2 weeks prior to the first dose of study drug.
17. Other exclusion criteria per protocol.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events of INBRX-109 | Up to 8 years
  Adverse events will be assessed and severity assigned by using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Evaluating Tumor Response for colorectal cancers and Ewing sarcoma | Up to 8 years
  Evaluating how the tumor responds to treatment by measuring the number of patients with colorectal cancer and Ewing sarcoma that experience tumor shrinkage and for how long.

SECONDARY OUTCOMES:
Immunogenicity of INBRX-109 | Up to 8 years
  Frequency of ant-drug antibodies (ADA) against INBRX-109 will be determined.
Characterize the pharmacokinetics of INBRX-109 as a single agent, and of INBRX-109 in combination with distinct chemotherapies. | Up to 8 years
  A measurement which indicates how the body processes INBRX-109 and how long it stays in the system.
Median progression-free survival for colorectal adenocarcinoma and Ewing sarcoma. | Up to 8 years
  Progression-free survival is defined as the time from start of study treatment until documented disease progression or death.

OTHER OUTCOMES:
Anti-tumor activity of INBRX-109 | Up to 8 years
  Tumor response will be determined by RECISTv1.1.
Potential predictive response biomarkers | Up to 8 years
  Evaluate the relationship between potential predictive response biomarkers and efficacy of INBRX-109

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Study Director — Inhibrx Biosciences, Inc
Locations (35):
- United States (22):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Precision NextGen Oncology and Research, Beverly Hills, California
  - City of Hope, Duarte, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of California, San Diego (UCSD) - Moores Cancer Center, San Diego, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Colorado Hospital, Aurora, Colorado
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - START Midwest Michigan, PC, Grand Rapids, Michigan
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia- Center for Childhood Cancer Research, Philadelphia, Pennsylvania
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - UT MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - NEXT Oncology - Virginia, Fairfax, Virginia
- France (2):
  - Centre Leon Berard, Lyon
  - Gustave Roussy, Villejuif
- Italy (2):
  - La Fondazione e l'Istituto di Candiolo, Candiolo
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Academisch Ziekenhuis Leiden, Leiden
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinico San Carlos, Madrid
- United Kingdom (4):
  - Great North Children's Hospital, London
  - University College London Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Subbiah V, Chawla SP, Conley AP, Wilky BA, Tolcher A, Lakhani NJ, Berz D, Andrianov V, Crago W, Holcomb M, Hussain A, Veldstra C, Kalabus J, O'Neill B, Senne L, Rowell E, Heidt AB, Willis KM, Eckelman BP. Preclinical Characterization and Phase I Trial Results of INBRX-109, A Third-Generation, Recombinant, Humanized, Death Receptor 5 Agonist Antibody, in Chondrosarcoma. Clin Cancer Res. 2023 Aug 15;29(16):2988-3003. doi: 10.1158/1078-0432.CCR-23-0974. PMID 37265425